CLINICAL TRIAL: NCT02851836
Title: Validation of an Attachment Picture Set in School-adolescent
Brief Title: Attachment Image Data Set Validation in Adolescent
Acronym: MONRADO1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: P/2012/152
Record Dates: First submitted 2016-07-26; First posted 2016-08-02 (Estimated); Last update posted 2016-08-02 (Estimated); Status verified 2016-07

CONDITIONS: Emotion Dysregulation
Keywords: attachment; adolescent; picture

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: image visualization and quotation — two sets of 60 pictures are shown to the adolescents. we ask them to quote for their valence, hedonicity, arousal and to characterize the emotion elicited in each picture.
  This evaluation takes approximately 1hour.

SUMMARY:
this study aims to validate a picture data set that particularly activates the attachment process and that could be used in attachment studies.

DETAILED DESCRIPTION:
Pictures have been chosen to represent several emotions: distress, comfort, complicity and neutral.

ELIGIBILITY:
Inclusion Criteria:

* adolescent going to high school not hospitalized

Exclusion Criteria:

* mental retardation non comprehension of french visual deficit

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 133 (Actual)
Dates: Start 2012-10; Primary Completion 2013-05 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
mean score of valence in the SAM (self assessment manikin system) | at inclusion
  the hedonicity is assessed for each picture. The characterization of the set is performed using the mean score of hedonicity for each type of picture (distress, comfort, complicity and neural)

SECONDARY OUTCOMES:
mean score of arousal in the SAM (self assessment manikin system) | at inclusion
  the hedonicity is assessed for each picture. The characterization of the set is performed using the mean score of arousal for each type of picture (distress, comfort, complicity and neural)
mean score of dominance in the SAM (self assessment manikin system) | at inclusion
  the hedonicity is assessed for each picture. The characterization of the set is performed using the mean score of dominance for each type of picture (distress, comfort, complicity and neural)
emotional categorization of the picture | at inclusion
  continuous scales for different emotions (distress, comfort, joy-complicity hate, horror) are presented. Subjects have to quote them for each picture.

CONTACTS AND LOCATIONS:
Overall Officials: Lauriane Vulliez-Coady, MD PhD, Principal Investigator — Centre Hospitalier Universitaire de Besancon
Locations (1):
- CHU Besancon, Besançon, Doubs, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Szymanska M, Monnin J, Noiret N, Tio G, Galdon L, Laurent E, Nezelof S, Vulliez-Coady L. The Besancon Affective Picture Set-Adolescents (the BAPS-Ado): Development and validation. Psychiatry Res. 2015 Aug 30;228(3):576-84. doi: 10.1016/j.psychres.2015.04.055. Epub 2015 Jun 20. PMID 26163722